CLINICAL TRIAL: NCT03053817
Title: The Impact of Structured Exercise on Brain Health in HIV Positive Individuals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Université du Québec a Montréal (Other)
Responsible Party: Principal Investigator, Nancy Mayo, Dr., McGill University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-384-MUHC
Record Dates: First submitted 2017-01-20; First posted 2017-02-15 (Actual); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: HIV

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise group (Experimental): The 45 minute exercise program will be performed 3 times a week and will consist of aerobic exercise and resistance training for 12 weeks.
  Interventions: Other: Exercise group
- Control (No Intervention): No treatment

INTERVENTIONS:
Other: Exercise group — Interval training will be performed for 21 minutes including a 3 minute warm-up and cool-down period. The interval program will be 15 minutes at 65-75% of maximal heart rate with 30 sec. bursts of exercise to 80-85%; intervals. Resistance training will be done as a circuit and will make use of weight machines and functional exercises. Resistance will be done in 2 sets of 15 repetitions and will last 24 minutes. The work load of the program is calibrated and is conducted at a specified rhythm. All exercise sessions will be supervised.
  Arms: Exercise group

SUMMARY:
Exercise programs that combine resistance exercise with aerobic training yield optimal health benefits for people with HIV. The global aim of this study is to contribute evidence for the impact potential of a comprehensive exercise program on brain health in people with HIV.

This study is part of a larger project based upon a cohort multiple randomized controlled design. Within a fully characterized cohort which is followed over time, people meeting the specific criteria for an exercise intervention will be identified. The sample will be randomly selected to receive the intervention; the remaining eligible persons will serve as controls. The intervention group will receive a 45 minute structured exercise program 3 times a week consisting of aerobic exercise and resistance training for a total of 12 weeks.

DETAILED DESCRIPTION:
Exercise is an inexpensive intervention with widespread benefits to vascular and musculoskeletal health and few harms. Showing an additional benefit to brain health and cognition in particular is likely to encourage adoption and help elucidate mechanisms underpinning brain health in HIV.

The primary objective of the study is to estimate, in comparison to individuals not offered the exercise intervention, the extent to which a comprehensive exercise program impacts on indicators of brain health, where these indicators are the primary outcome of cognitive ability (B-CAM) and the related brain health outcomes of depression, anxiety, fatigue, motivation, and speed of motor performance.

A secondary objective is to estimate the extent to which changes in brain health are mediated through exercise induced changes in brain network function as measured by EEG and/or by exercise induced changes in muscle power, aerobic capacity, physical function, and body composition.

ELIGIBILITY:
The exercise intervention will target individuals recruited from two Montreal clinics who identified at cohort entry they were interested in being approached for different trials if they eligible.

Inclusion Criteria:

* men and women aged ≥ 35 years, HIV+ for at least 1 year, able to communicate adequately in either French or English, and able to give written informed consent.

Also, participants must identify that they are mostly sedentary by reporting that they perform moderate level physical activity of 30 minutes duration less than twice a week or have limitations in performing vigorous activities, walking a kilometer, or climbing stairs. Individuals answering yes to any of the Physical Activities Readiness Questionnaire (PAR-Q) (Thomas et al., 1992) items except taking medication (Item 6) will require clearance from their physician to be included.

Exclusion Criteria:

* people with dementia (MOCA < 18) or treating physician's concern about capacity to consent, life expectancy of < 3 years or other personal factors limiting the ability to participate in follow-up, non-HIV-related neurological disorder likely to affect cognition, known active CNS opportunistic infection or hepatitis C requiring interferon (IFN) treatment during the follow-up period, psychiatric disorder on the psychotic axis, current substance use disorder or severe substance use disorder within the past 12 months.

Also excluded will be people with a contraindication for exercise from cardiovascular or musculoskeletal co-morbidity as gathered from the medical history and from the PAR-Q (Thomas et al., 1992).

Ages: 35 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-12; Primary Completion 2018-01 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in Cognitive Ability | 0 and 39 weeks
  The primary outcome is cognitive ability as measured by B-CAM. This is part of the measurement platform for all and the value taken at the regular assessment prior to the exercise intervention will serve as the baseline value and the subsequent evaluation 9 months following will serve as the follow-up value. The strategy ensures that the intervention cohort does not have additional measurements of cognitive ability than the control cohort. The items on the B-CAM fit the Rasch Model and as such have linearized units on a logit scale.

SECONDARY OUTCOMES:
Change in depression | 0 and 39 weeks
  Measured by Hospital Anxiety and Depression Scale (HADS)
Change in depression | 0 and 39 weeks
  Measured by RAND -36 Mental Health Inventory (MHI)
Change in stress levels | 0 and 39 weeks
  Measured by Trier Inventory for Chronic Stress (TICS)
Change in anxiety | 0 and 39 weeks
  Measured by Hospital Anxiety and Depression Scale (HADS)
Change in fatigue | 0 and 39 weeks
  Measured by RAND-36 Vitality
Change in motivation | 0 and 39 weeks
  Measured by Motivation Ladder
Change in global quality of life (QOL) | 0 and 39 weeks
  Measured by Person Generated Index (PGI)
Change in health related quality of life (HRQoL) | 0 and 39 weeks
  Measured by RAND-36
Change in health related quality of life (HRQoL) | 0 and 39 weeks
  Measured by WHOQOL-HIV
Change in measures of brain network function | 0 and 12 weeks
  The measures of brain network function are derived from event related potential (ERPs) which are electric potentials produced by the brain in response to auditory or visual stimulation, respectively. These brain responses are easily recorded noninvasively with scalp electrodes (EEG). ERPs allow insights into the neural mechanisms underlying specific cognitive processes. The potentials of interest here include the N1, N2, P2 and P3 ERPs.
Change in skeletal muscle mass | 0 and 12 weeks
  A total body Dual energy X-ray absorptiometry (DEXA) scan will be done to compute skeletal muscle mass (whole body, spine and thigh) (Lee & Gallagher, 2009).
Change in muscle quality | 0 and 12 weeks
  Peripheral quantitative computed tomography (pQCT) will be used to measure the muscle quality in lower extremity (MacIntyre & Lorbergs, 2012).
Change in exercise capacity | 0 and 12 weeks
  Measured by step test
Change in functional walking capacity | 0 and 12 weeks
  Measured by Six Minute Walk Test (6MWT)
Change in quadriceps power | 0 and 12 weeks
  Measured using leg press and jump test
Change in core strength | 0 and 12 weeks
  Measured using curl ups/push ups
Change in grip strength | 0 and 12 weeks
  Measured using hand dynamometer
Change in gait speed | 0 and 12 weeks
  Comfortable gait speed: GAITRite; Fast gait speed: GAITRite; Dual task gait speed: GAITRite and naming the fruits
Change in exercise enjoyment | 0 and 12 weeks
  Exercise enjoyment will be measured by Physical Activity Enjoyment Scale (PACES) (Mullen et al., 2011).
Change in physical activity | 0, 6 and 12 weeks
  The data from the accelerometer will be used to estimate the extent to which the structured exercise program carries over into everyday life. Participants will be asked to wear an ActivPal accelerometer for 5-7 days prior to the start of the intervention, at 6 weeks, and after 12 weeks, to objectively measure habitual physical activity.
Change in semantic fluency | 0 and 12 weeks
  Following question will be asked:
  Name as many animals as you can in 1 minute (in sitting).

CONTACTS AND LOCATIONS:
Overall Officials: Nancy E Mayo, PhD, Principal Investigator — McGill University
Locations (1):
- Division of Clinical Epidemiology, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Relton C, Torgerson D, O'Cathain A, Nicholl J. Rethinking pragmatic randomised controlled trials: introducing the "cohort multiple randomised controlled trial" design. BMJ. 2010 Mar 19;340:c1066. doi: 10.1136/bmj.c1066. No abstract available. PMID 20304934
- [Background] Mullen SP, Olson EA, Phillips SM, Szabo AN, Wojcicki TR, Mailey EL, Gothe NP, Fanning JT, Kramer AF, McAuley E. Measuring enjoyment of physical activity in older adults: invariance of the physical activity enjoyment scale (paces) across groups and time. Int J Behav Nutr Phys Act. 2011 Sep 27;8:103. doi: 10.1186/1479-5868-8-103. PMID 21951520
- [Background] Lee SY, Gallagher D. Assessment methods in human body composition. Curr Opin Clin Nutr Metab Care. 2008 Sep;11(5):566-72. doi: 10.1097/MCO.0b013e32830b5f23. PMID 18685451
- [Background] Macintyre NJ, Lorbergs AL. Imaging-Based Methods for Non-invasive Assessment of Bone Properties Influenced by Mechanical Loading. Physiother Can. 2012 Spring;64(2):202-15. doi: 10.3138/ptc.2011-08bh. Epub 2012 Apr 5. PMID 23449969
- [Background] Thomas S, Reading J, Shephard RJ. Revision of the Physical Activity Readiness Questionnaire (PAR-Q). Can J Sport Sci. 1992 Dec;17(4):338-45. PMID 1330274
- [Background] Malita FM, Karelis AD, Toma E, Rabasa-Lhoret R. Effects of different types of exercise on body composition and fat distribution in HIV-infected patients: a brief review. Can J Appl Physiol. 2005 Apr;30(2):233-45. doi: 10.1139/h05-117. PMID 15981790